CLINICAL TRIAL: NCT03229252
Title: A Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy and Safety of SPX-101 Inhalation Solution in Subjects With Cystic Fibrosis (HOPE-1 Study: Hydration for Optimal Pulmonary Effectiveness)
Brief Title: An Efficacy and Safety Study of SPX-101 Inhalation Solution in Subjects With Cystic Fibrosis
Acronym: (HOPE-1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spyryx Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPX-101-CF-201
Record Dates: First submitted 2017-07-14; First posted 2017-07-25 (Actual); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo Inhalation solution twice daily for 28 days.
  Interventions: Drug: Placebo Inhalation Solution
- SPX-101 Low Dose (Experimental): Inhalation solution twice daily for 28 days.
  Interventions: Drug: SPX-101
- SPX-101 High Dose (Experimental): Inhalation solution twice daily for 28 days.
  Interventions: Drug: SPX-101

INTERVENTIONS:
Drug: Placebo Inhalation Solution — Normal Saline Inhalation Solution
  Arms: Placebo
Drug: SPX-101 — SPX-101 Inhalation Solution
  Arms: SPX-101 High Dose; SPX-101 Low Dose

SUMMARY:
28-Day double-blinded efficacy and safety trial of SPX-101 Inhalation Solution in adult subjects with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cystic fibrosis
* ppFEV1 (percent predicted FEV1) between 50.0% and 80.0%
* Stable CF Lung Disease
* Males and non-pregnant, non-lactating females

Exclusion Criteria:

* Significant unstable co-morbidities within 28 days of screening
* Has received an investigational drug within 28 days of screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- Canada (3):
  - University of Calgary Heritage Medical Research Center, Calgary, Alberta
  - Ottawa Hospital Research Institute/Institut de Recherche de l'Hospital d'Ottawa, Ottawa, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
- France (7):
  - Hospices Civils de Lyon (HCL), Pierre-Bénite, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire Brest, Roscoff, Brittany Region
  - CHU de Rouen, Rouen, Haute-Normandie
  - CHU de Montpellier, Montpellier, Languedoc-Roussillon
  - CHU de Angers, Angers, Pays de la Loire Region
  - Hopital Pasteur, Nice, Provence-Alpes-Côte d'Azur Region
  - Assistance Publique-Hôpitaux de Paris Hôpital Cochin, Paris
- Istituto Giannina Gaslini Ospedale Pediatrico, Genoa, Italy
- Hospital de Santa Maria, Lisbon, Portugal
- United Kingdom (13):
  - Belfast Health and Social Care Trust, Belfast
  - Heart of England NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Western General Hospital - NHS Lothian, Edinburgh
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - NHS Greater Glasgow and Clyde, Glasgow
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust Saint Bartholomews Hospital, London
  - Royal Brompton and Harefield NHS Foundation Trust, London
  - University Hospital of South Manchester NHS Foundation Trust, Manchester
  - Newcastle Upon Tyne Hospitals, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SPX-101 Low Dose (60mg BID); SPX-101 High Dose (120mg BID): Inhalation solution twice daily for 28 days.
  SPX-101: SPX-101 Inhalation Solution
Period: Overall Study
Arm/Group | Placebo | SPX-101 Low Dose (60mg BID) | SPX-101 High Dose (120mg BID)
Started | 31 | 15 | 45
Completed | 29 | 15 | 39
Not Completed | 2 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SPX-101 Low Dose (60mg BID) | SPX-101 High Dose (120mg BID) | Total
Number analyzed (Participants) | 31 | 15 | 45 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 15 | 45 | 91
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (7.82) | 33.7 (8.62) | 31.9 (8.49) | 31.8 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 22 | 37
  Male | 20 | 11 | 23 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 29 | 14 | 43 | 86
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 26 | 12 | 44 | 82
  More than one race | 3 | 3 | 1 | 7
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 5 | 8 | 16
  Italy | 1 | 0 | 3 | 4
  United Kingdom | 14 | 7 | 15 | 36
  France | 12 | 2 | 13 | 27
  Portugal | 1 | 1 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Predicted FEV1
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: change from baseline in ppFEV1
Arm/Group | Placebo | SPX-101 Low Dose (60mg BID) | SPX-101 High Dose (120mg BID)
Number analyzed (Participants) | 31 | 15 | 45
change from baseline in ppFEV1 | 1.633 (6.3302) | 0.800 (6.5049) | 0.890 (6.7061)

2. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Day 1 through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SPX-101 Low Dose (60mg BID) | SPX-101 High Dose (120mg BID)
Number analyzed (Participants) | 31 | 15 | 45
Participants | 20 | 11 | 30

3. Secondary Outcome: Change From Baseline Through Day 28 in Clinical Laboratory Tests
Description: Chemistry, Hematology, Urinalysis
Time Frame: Day 1 through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SPX-101 Low Dose (60mg BID) | SPX-101 High Dose (120mg BID)
Number analyzed (Participants) | 31 | 15 | 45
Participants
  Blood Electrolytes (Potassium) Low | 0 | 0 | 0
  Blood Electrolytes (Potassium) Normal | 29 | 13 | 40
  Blood Electrolytes (Potassium) High | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 28 Days
Arm/Group | Placebo | SPX-101 Low Dose (60mg BID) | SPX-101 High Dose (120mg BID)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/15 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/15 | 3/45
Other Adverse Events (participants affected / at risk) | 20/31 | 10/15 | 29/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | SPX-101 Low Dose (60mg BID) (N=15) | SPX-101 High Dose (120mg BID) (N=45)
Infective Pulmonary Exacerbation of Cystic Fibrosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intestinal Obstuction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough and Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | SPX-101 Low Dose (60mg BID) (N=15) | SPX-101 High Dose (120mg BID) (N=45)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 6 (6)
Sputum Increased (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 4 (7)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Lower Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Increased Viscosity of Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sputum Discolored (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infective Pulmonary Exacerbation of Cystic Fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (3)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue Coated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 2 (2) | 2 (2) | 2 (3)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Forced Expiratory Volume Decreased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
No Limitations or Caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT03229252/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT03229252/SAP_001.pdf